CLINICAL TRIAL: NCT04646174
Title: Addressing Psychological Risk Factors Underlying Smoking Persistence: The Fresh Start-II Study
Brief Title: Addressing Psychological Risk Factors Underlying Smoking Persistence in COPD Patients: The Fresh Start-II Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18082201
Record Dates: First submitted 2020-11-20; First posted 2020-11-27 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Copd; Smoking Cessation; Nicotine Dependence; Tobacco Use; Cigarette Smoking
Keywords: Copd; Smoking Cessation; Nicotine Dependence; Tobacco Use; Cigarette Smoking; Behavioral Treatment; Self-guided Treatment
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking Cessation; Tobacco Use Disorder; Tobacco Use; Cigarette Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-component Behavioral Treatment (Experimental): This treatment consists of nine weekly phone-based individual treatment sessions, 45-60 minutes each, delivered by a trained study therapist.
  Interventions: Behavioral: Unified Protocol adapted for smoking cessation; Behavioral: American Lung Association self-management strategies for smoking cessation
- Self-guided Treatment (Experimental): This treatment consists of self-help materials from the American Lung Association that address evidence-based smoking cessation and self-management strategies.
  Interventions: Behavioral: American Lung Association self-management strategies for smoking cessation

INTERVENTIONS:
Behavioral: Unified Protocol adapted for smoking cessation — Treatment components are cognitive-behavioral strategies adapted from the Unified Protocol (UP) for the Transdiagnostic Treatment of Emotional Disorders. Behavioral counseling strategies for smoking cessation, drawn from current US Public Health Service guidelines, are incorporated in each treatment module.
  Arms: Multi-component Behavioral Treatment
Behavioral: American Lung Association self-management strategies for smoking cessation — Treatment components are self-management strategies provided through printed self-help materials from the American Lung Association. The materials consist of the Freedom from Smoking guide, Relaxation Exercises for Better Breathing, and COPD; Exercise and Daily Activity guide that address evidence-based smoking cessation and self-management strategies to aid in a quit attempt.

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is caused primarily by smoking and smoking cessation is the first-line treatment for slowing disease progression. Despite this, nearly 50% of COPD patients continue to smoke following diagnosis. Smokers with COPD report high rates of co-occurring conditions - nicotine dependence, depression, and anxiety - which serve as barriers to quitting. The current study will pilot test a behavioral intervention designed to target the common psychological factors underlying these co-occurring conditions and foster smoking cessation among COPD patients.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is caused primarily by smoking and smoking cessation is the first-line treatment for slowing disease progression. Despite this, nearly 50% of COPD patients continue to smoke following diagnosis. Smokers with COPD report high rates of co-occurring conditions - nicotine dependence, depression, and anxiety - which serve as barriers to quitting. The proposed research will develop and pilot test a behavioral intervention designed to target the common psychological factors underlying these co-occurring conditions and foster smoking cessation among COPD patients. The specific aim is to:

Aim: Examine effects of psychological risk factor reduction on smoking outcome. We will conduct a pilot trial in which 62 participants are randomized to the multi-component behavioral treatment (9 weekly sessions) or self-guided treatment (mailing of printed self-help materials).The primary outcome is number of days abstinent for 2 weeks post-quit (range = 0-14 days).

ELIGIBILITY:
Inclusion Criteria:

Eligible participants will be males and females who are:

* Diagnosed with COPD (as documented in electronic health record [EHR]),
* Daily cigarette smokers (5 or more cigarettes per day over past 30 days),
* Intend to quit smoking within the next 60 days,
* Report at least moderate level of smoking for affective regulation (SMQ-R coping subscale score 30 or greater),
* Have access to a smart phone, tablet, or computer, and
* Are able to communicate fluently in English

Exclusion Criteria:

* Any concurrent medical or psychiatric condition which would preclude ability to provide informed consent or perform study procedures (e.g., moderate to severe dementia and/or severe, uncontrolled schizophrenia), as determined by the treating physician or study PI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Two-Week Smoking Abstinence | 14 days post-quit date
  Number of days abstinent for 2 weeks post-quit, as verified by CO < 5 ppm

SECONDARY OUTCOMES:
Smoking Status | 3 months post-quit
  Self-reported 7-day point prevalence abstinence, as verified by CO < 5 ppm

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Mathew, PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No